CLINICAL TRIAL: NCT02197039
Title: The Selection Criteria for Deciding Who Needs the Second-look Endoscopy Among Patients With Bleeding Peptic Ulcers
Brief Title: The Selection Criteria for the Second-look Endoscopy Among Patients With Bleeding Peptic Ulcers
Acronym: CSE
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: A-ER-103-112
Record Dates: First submitted 2014-07-20; First posted 2014-07-22 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2014-07

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: Peptic ulcer hemorrhage, second-look endoscopy
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — Esomeprazole; Pantoprazole; Hemostasis, Endoscopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, gastric tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- The High risk group: Each enrolled patient receives an 80 mg loading dose of intravenous esomeprazole or pantoprazole immediately after successful endoscopic hemostasis. Patients then receive a 3-day continuous high dose (8 mg per hour) of esomeprazole or pantoprazole infusion.
  Patients are defined in the high risk group if they still have major stigmata of recent hemorrhage at the second-look endoscopy or have early recurrent bleeding before the schedule time for follow-up.
  Recurrent bleeding is defined as: 1) continuous melena, hematochezia, or the presence of recurrent bloody aspirates through a nasogastric tube and 2) relapse of hemodynamic instability, including systolic blood pressure <90 mmHg, heart rate >120 beats per minute, or a drop in hemoglobin concentration by more than 2 g/dL.
  Interventions: Drug: esomeprazole or pantoprazole; Procedure: Endoscopic hemostasis
- The control group: Each enrolled patient receives an 80 mg loading dose of intravenous esomeprazole or pantoprazole immediately after successful endoscopic hemostasis. Patients then receive a 3-day continuous high dose (8 mg per hour) of esomeprazole or pantoprazole infusion.
  Patients are defined in the control group if they does not have recurrent bleeding before the schedule time for follow-up, and have only minor stigmata of hemorrhage or clean ulcer base at the second-look endoscopy.
  Recurrent bleeding is defined as: 1) continuous melena, hematochezia, or the presence of recurrent bloody aspirates through a nasogastric tube and 2) relapse of hemodynamic instability, including systolic blood pressure <90 mmHg, heart rate >120 beats per minute, or a drop in hemoglobin concentration by more than 2 g/dL.
  Interventions: Drug: esomeprazole or pantoprazole; Procedure: Endoscopic hemostasis

INTERVENTIONS:
Drug: esomeprazole or pantoprazole — Each enrolled patient receives an 80 mg loading dose of intravenous esomeprazole (Nexium®, AstraZeneca AB, Södertälje, Sweden) immediately after hemostasis is achieved spontaneously or by gastroscopy. Patients then receive a 3-day continuous high dose (8 mg per hour) of esomeprazole infusion. Because of concern for patient safety with certain drug-drug interactions, patients who take clopidogrel receive intravenous pantoprazole (Pantoloc®, Takeda, Singen, Germany), including an 80 mg loading dose and a 3-day continuous high-dose (8 mg/h) of infusion.
  Other Names: Nexium® (AstraZeneca AB) or Pantoloc® (Takeda)
Procedure: Endoscopic hemostasis — At the index gastroscopy, bleeding ulcers are checked. If the adherent clot is found over the ulcer base, it will be vigorously washed away with water jet. All of the stigmata of recent hemorrhage (SRH) are treated by one or a combination of endoscopic therapies including local injection of diluted epinephrine 1:10000, bipolar heated probe at 20 J per goal consecutively until achievement of coaptive coagulation, argon plasma coagulation, band ligation, or hemoclip therapy. The success of endoscopic hemostasis is defined as cessation of bleeding together with achievement of cavitation at the vessel after application of the heater probe.

SUMMARY:
The purpose of this prospective study is to identify risk factors which could predict poor fading of SRH or early recurrent bleeding of peptic ulcer hemorrhage after successful endoscopic hemostasis and high-dose PPI infusion. These risk factors will be the selection criteria for patients who are indicated to receive second-look endoscopy.

DETAILED DESCRIPTION:
Peptic ulcer bleeding is a common disease, and recurrent bleeding is an independent risk factor leading to mortality. The appearance of stigmata of recent hemorrhage (SRH) indicates possible recurrence of peptic ulcer bleeding, for which the likelihood decreases over the course of 3-6 days. In addition to endoscopic evidences illustrating the SRH, patients with co-morbidities have a higher risk of recurrent bleeding.

Patients with co-morbidities have not only higher recurrent bleeding rates during the first 3 days but also higher delay recurrent bleeding after 3-day proton pump inhibitor (PPI) infusion than those without. More than 50% recurrent bleeding develops after 3-day PPI infusion among patients with end stage renal diseases. Although endoscopic treatment plus a 72-hour intravenous PPI infusion and followed by oral PPI has already been adopted as a standard treatment in peptic ulcer bleeding currently, several studies showed limited effectiveness of such treatment for high risk patients. The reasons may be because lesions of SRH were not completely faded after initial treatment including endoscopic hemostasis and intravenous PPI infusion. Thus, it is an important issue to improve such high recurrent bleeding risk for these patients.

Endoscopic treatment plus a 72-hour intravenous PPI infusion is the standard protocol for treatment of peptic ulcer bleeding. Moreover, several studies have shown that PPI treatment could decrease the presentation of SRH. However, there were insufficient data to validate the efficacy of such standard treatment to fade the SRH, especially among high risk patients. Therefore, several studies looked at the efficacy of routine second-look endoscopy, defined as scheduled repeat endoscopy after primary endoscopic hemostasis in patients at high risk of rebleeding. However, the role and the selection criteria for patients who require second-look endoscopy remains uncertain. There is a pressing need to elucidate the role of second-look endoscopy in these patients.

Hence, the purpose of this prospective study is to identify risk factors which could predict poor fading of SRH or early recurrent bleeding of peptic ulcer hemorrhage after successful endoscopic hemostasis and high-dose PPI infusion. This data will show the originality and clinical importance to identify the selection criteria for patients who are indicated to receive second-look endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Bleeding peptic ulcers with major stigmata of recent hemorrhage
* All of these major SRH are treated by local injection of diluted epinephrine 1:10000 with or without combined therapy with a heater probe, argon plasma coagulation, band ligation, or hemoclip therapy

Exclusion Criteria:

* Bleeding due to tumor or cancer
* Bleeding due to the presence of a Dieulafoy lesion
* Ulcer bleeding due to mechanical factors (i.e., gastrostomy tube induction)
* Proton pump inhibitors use within one week before enrollment
* Failure to establish hemostasis under gastroscopy
* Hypersensitivity to esomeprazole, pantoprazole, or any component of the formulation
* Previously participated in the study

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We developed the study with data collected in an audit of admissions for acute peptic ulcer hemorrhage at the inpatient wards of National Cheng Kung University Hospital, a tertiary health care center in Tainan, Taiwan. Patients who receive gastroscopy for melena, hematochezia, or hematemesis in whom bleeding peptic ulcers with major stigmata of recent hemorrhage are detected are consecutively enrolled.
Sampling Method: Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2011-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
the fading rate of major stigmata of recent hemorrhage | within 3 days after the index gastroscopy
  At the index gastroscopy, bleeding ulcers are checked. All of the major stigmata of recent hemorrhage (SRH) are treated by one or a combination of endoscopic therapies. The success of endoscopic hemostasis is defined as cessation of bleeding together with achievement of cavitation at the vessel after application of the heater probe.
  Second-look endoscopy is scheduled 48-72 hours after successful index endoscopic hemostasis and intravenous high-dose proton pump inhibitor infusion. For each patient with either suspected or active recurrent bleeding, emergent endoscopy is conducted earlier before the schedule to confirm peptic ulcer recurrent bleeding.
  Possible risk factors including patient's baseline clinical, laboratory characteristics, and gastroscopic pictures are obtained at the time of admission.
  Multiple logistic regression analysis is applied to assess the independent risk factors related to residual major stigmata or early recurrent bleeding of peptic ulcers.

CONTACTS AND LOCATIONS:
Overall Officials: Bor-Shyang Sheu, MD, Study Director — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Derived] Cheng HC, Wu CT, Chen WY, Yang EH, Chen PJ, Sheu BS. Risk factors determining the need for second-look endoscopy for peptic ulcer bleeding after endoscopic hemostasis and proton pump inhibitor infusion. Endosc Int Open. 2016 Mar;4(3):E255-62. doi: 10.1055/s-0041-111499. Epub 2016 Feb 8. PMID 27004241